CLINICAL TRIAL: NCT02013934
Title: Benefit and Tolerability of a Probiotic Product in Subjects With Increased Susceptibility to Common Cold
Brief Title: Probiotics in Prevention of Common Cold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PAB/011013
Record Dates: First submitted 2013-12-06; First posted 2013-12-17 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2013-12

CONDITIONS: Viral Infections of the Upper Respiratory Tract
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics (Active Comparator): Dietary supplement
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Dietary supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic
  Arms: Probiotics
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the benefit and tolerability of a probiotic product in subjects with increased susceptibility to common cold.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* age 18-70 years
* increased risk for common cold (at least 4 episodes within 12 months)
* commitment to adhere to former diet and physical activity
* commitment not to use any products that may influence the study outcome (e.g. immune suppressants/immune stimulants, including paramedication such as e.g. Echinacea, analgesics/anti-rheumatics, anti-phlogistics, antitussives/expectorants, influenza remedies, mouth or throat therapeutics, decongestants, antibiotics, anti-histaminergic drugs, probiotics) during the study (except for rescue medication, see 7.5)
* women of child-bearing potential have to agree to use appropriate birth control methods Written consent of the subject to participate is a prerequisite for study participation.

Exclusion Criteria:

* acute / chronic upper / lower airways disease
* chronic cough of any origin
* any allergic reaction that may influence the study outcome (e.g. acute/chronic rhinitis)
* history of nasal reconstructive surgery
* presence of nasal ulcers or nasal polyps
* severe nasal septum deviation or other condition that could cause nasal obstruction
* congenital or acquired immunodeficiency disease (e.g. HIV infection)
* Bechterew's disease
* body temperature above 37.5°C
* suspected swine flu or influenza
* vaccination with a vaccine containing an adjuvant within 3 months prior to study start and during the study
* vaccination with a vaccine not containing an adjuvant within 6 weeks prior to study start and during the study
* stomach/gastrointestinal diseases
* serious organ or systemic diseases
* sleep disorder
* psychiatric disorders
* known sensitivity to the ingredients of the investigational product
* regular intake of products that may influence the study outcome (e.g. immune suppressants/immune stimulants, including paramedication such as e.g. Echinacea, analgesics/anti-rheumatics, anti-phlogistics, antitussives/expectorants, influenza remedies, mouth or throat therapeutics, decongestants, antibiotics, anti-histaminergic drugs, probiotics) within the last 4 weeks prior to study start
* habitual usage of nasal drops/spray
* pregnancy or nursing
* alcohol / drug abuse
* simultaneous participation in another clinical trial or participation in a clinical trial within the last 30 days
* insufficient compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 899 (Actual)
Dates: Start 2013-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05-17 (Actual)

PRIMARY OUTCOMES:
Severity of cold symptoms | 3 months
  Severity of cold symptoms based on the questionnaire WURSS-21 during the cold episodes throughout the study period, in comparison between verum and placebo group

SECONDARY OUTCOMES:
Incidence of common cold episodes | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- A&R, Berlin, Germany

REFERENCES:
- [Derived] Ahren IL, Hillman M, Nordstrom EA, Larsson N, Niskanen TM. Fewer Community-Acquired Colds with Daily Consumption of Lactiplantibacillus plantarum HEAL9 and Lacticaseibacillus paracasei 8700:2. A Randomized, Placebo-Controlled Clinical Trial. J Nutr. 2021 Jan 4;151(1):214-222. doi: 10.1093/jn/nxaa353. PMID 33296464